CLINICAL TRIAL: NCT04177693
Title: Pharmacokinetics and Hepatic Safety of EGCG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Illinois at Chicago (Other); Johns Hopkins University (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Hugh Taylor, Chair of Obstetrics, Gynecology and Reproductive Sciences, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000028370; 1R01HD100369-01 (NIH)
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — epigallocatechin gallate; Clomiphene; Letrozole

STUDY DESIGN:
Intervention Model Description: The 36 women will be randomized to one of the following groups:
  1. EGCG daily alone.
  2. EGCG daily with clomiphene citrate 100mg for 5 days.
  3. EGCG daily with letrozole 5mg for 5 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EGCG daily alone. (Experimental): EGCG daily alone. 800mg
  Interventions: Dietary Supplement: Epigallocatechin gallate (EGCG)
- EGCG with clomiphene citrate (Experimental): EGCG 800 mg daily with clomiphene citrate 100mg for 5 days.
  Interventions: Dietary Supplement: Epigallocatechin gallate (EGCG); Drug: Clomiphene Citrate
- EGCG with letrozole (Experimental): EGCG 800mg daily with letrozole 5mg for 5 days.
  Interventions: Dietary Supplement: Epigallocatechin gallate (EGCG); Drug: Letrozole

INTERVENTIONS:
Dietary Supplement: Epigallocatechin gallate (EGCG) — 800 mg (4 capsules) of EGCG (green tea extract), taken orally on a daily basis for up to 2 months
Drug: Clomiphene Citrate — 100 mg for 5 days
  Other Names: Clomid; Serophene
  Arms: EGCG with clomiphene citrate
Drug: Letrozole — 5 mg for 5 days
  Other Names: Femara
  Arms: EGCG with letrozole

SUMMARY:
A trial to assess the pharmacokinetics and hepatic safety of EGCG in women with and without uterine fibroids.

DETAILED DESCRIPTION:
This will be a randomized, multi-center, pharmacokinetics and hepatic safety trial of EGCG with 36 total patients in 3 treatment arms. 36 women will be randomized to one of the following groups: EGCG daily alone, EGCG daily with clomiphene citrate and EGCG daily with letrozole. The randomization scheme will be stratified for age groups 18-29 and 30-40 and presence of uterine fibroids. The pharmacokinetics and hepatic safety of EGCG with clomiphene citrate and letrozole are unknown. The trial conducted in women with and without fibroids will allow comparisons between these groups. The results of this study will be used to confirm hepatic safety for the larger multi-center FRIEND study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women ≥18 to ≤40 years of age with or without uterine fibroids
2. Must use a double-barrier method for contraception

Exclusion Criteria:

1. Subjects using green tea/EGCG within 2 weeks prior to study enrollment
2. Known liver disease (defined as AST or ALT>2 times normal, or total bilirubin >2.5 mg/dL).
3. History of alcohol abuse (defined as >14 drinks/week) or binge drinking of ≥ 6 drinks at one time).
4. Subject using hormonal contraceptives
5. Subjects who are pregnant or breastfeeding
6. Known hypersensitivity to the study drugs
7. Any chronic disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Eisenberg, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Ayman Al-Hendy, MD,PhD, Principal Investigator — University of Chicago; Heping Zhang, PhD, Study Director — Yale University; James Segars, MD, Study Director — Johns Hopkins University; Hugh Taylor, MD, Study Director — Yale University; Frank Gonzales, MD, Study Director — University of Illinois Chicago
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EGCG Daily Alone. | EGCG With Clomiphene Citrate | EGCG With Letrozole
Started | 16 | 11 | 12
Completed | 14 | 11 | 11
Not Completed | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EGCG Daily Alone. | EGCG With Clomiphene Citrate | EGCG With Letrozole | Total
Number analyzed (Participants) | 16 | 11 | 12 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (6.3) | 27.2 (6.6) | 29.3 (6.3) | 28.8 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 12 | 39
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 14 | 9 | 10 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 2 | 2 | 1 | 5
  White | 11 | 6 | 6 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Changes in Epigallocatechin Gallate (EGCG)
Description: Changes in epigallocatechin gallate (EGCG) from Visit 1 to Visit 4 (end of study). EGCG levels measured at 1 hour after taking study medication were used for both visits.
Time Frame: Baseline, and Visit 4 (end of study, up to 40 days)
Measure: Median (Inter-Quartile Range); unit: nM
Arm/Group | EGCG Daily Alone. | EGCG With Clomiphene Citrate | EGCG With Letrozole
Number analyzed (Participants) | 12 | 10 | 8
nM | 5.8 [-418.2 to 263.1] | 256.3 [37.9 to 770.1] | 86.4 [-130.6 to 788.1]
Statistical Analysis 1: Comparison: EGCG Daily Alone. vs EGCG With Clomiphene Citrate vs EGCG With Letrozole; Test type: Superiority; p = 0.112, Kruskal-Wallis

2. Primary Outcome: Changes in Epigallocatechin (EGC)
Description: Changes in epigallocatechin (EGC) from Visit 1 to Visit 4 (end of study). EGC levels measured at 1 hour after taking study medication were used for both visits.
Time Frame: Baseline, and Visit 4 (end of study, up to 40 days)
Measure: Median (Full Range); unit: nM
Arm/Group | EGCG Daily Alone. | EGCG With Clomiphene Citrate | EGCG With Letrozole
Number analyzed (Participants) | 5 | 5 | 5
nM | -58.9 [-66.2 to 62.2] | 8.9 [-0.3 to 17.3] | 35.4 [-19.7 to 193.6]
Statistical Analysis 1: Comparison: EGCG Daily Alone. vs EGCG With Clomiphene Citrate vs EGCG With Letrozole; Test type: Superiority; p = 0.613, Kruskal-Wallis

3. Primary Outcome: Changes in Epicatechin Gallate(ECG)
Description: Changes in epicatechin gallate(ECG) from Visit 1 to Visit 4 (end of study). ECG levels measured at 1 hour after taking study medication were used for both visits.
Time Frame: Baseline, and Visit 4 (end of study, up to 40 days)
Measure: Median (Inter-Quartile Range); unit: nM
Arm/Group | EGCG Daily Alone. | EGCG With Clomiphene Citrate | EGCG With Letrozole
Number analyzed (Participants) | 10 | 5 | 9
nM | 7.6 [-121.7 to 63.0] | 64.1 [1.0 to 248.0] | 60.3 [-20.2 to 127.7]
Statistical Analysis 1: Comparison: EGCG Daily Alone. vs EGCG With Clomiphene Citrate vs EGCG With Letrozole; Test type: Superiority; p = 0.202, Kruskal-Wallis

4. Secondary Outcome: Changes in Total Bilirubin
Description: Changes in total bilirubin between the 3 groups.
Time Frame: Baseline, and Visit 4 (end of study, up to 40 days)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | EGCG Daily Alone. | EGCG With Clomiphene Citrate | EGCG With Letrozole
Number analyzed (Participants) | 15 | 11 | 12
mg/dL | 0.1 (0.2) | 0 (0) | 0 (0.1)
Statistical Analysis 1: Comparison: EGCG Daily Alone. vs EGCG With Clomiphene Citrate vs EGCG With Letrozole; Test type: Superiority; p = 0.508, Kruskal-Wallis

5. Secondary Outcome: Changes in ALT/SGPT
Description: Changes in alanine aminotransferase /SGPT between the 3 groups.
Time Frame: Baseline, and Visit 4 (end of study, up to 40 days)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | EGCG Daily Alone. | EGCG With Clomiphene Citrate | EGCG With Letrozole
Number analyzed (Participants) | 15 | 11 | 12
U/L | 1.1 (5.1) | 4.4 (11.7) | -1.0 (7.6)
Statistical Analysis 1: Comparison: EGCG Daily Alone. vs EGCG With Clomiphene Citrate vs EGCG With Letrozole; Test type: Superiority; p = 0.237, Kruskal-Wallis

6. Secondary Outcome: Changes in Alkaline Phosphatase
Description: Changes in Alkaline Phosphatase between the 3 groups.
Time Frame: Baseline, and Visit 4 (end of study, up to 40 days)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | EGCG Daily Alone. | EGCG With Clomiphene Citrate | EGCG With Letrozole
Number analyzed (Participants) | 15 | 11 | 12
U/L | -1.5 (5.4) | -5.6 (10.2) | -6.0 (9.1)
Statistical Analysis 1: Comparison: EGCG Daily Alone. vs EGCG With Clomiphene Citrate vs EGCG With Letrozole; Test type: Superiority; p = 0.327, Kruskal-Wallis

7. Secondary Outcome: Changes in Estrogen (E2)
Description: Changes in Estrogen (E2) between the 3 groups.
Time Frame: Baseline, and Visit 4 (end of study, up to 40 days)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | EGCG Daily Alone. | EGCG With Clomiphene Citrate | EGCG With Letrozole
Number analyzed (Participants) | 15 | 11 | 12
pg/mL | -50.9 (122.4) | -49.4 (76.6) | -50.2 (127.9)
Statistical Analysis 1: Comparison: EGCG Daily Alone. vs EGCG With Clomiphene Citrate vs EGCG With Letrozole; Test type: Superiority; p = 0.633, Kruskal-Wallis

8. Secondary Outcome: Changes in Endometrial Thickness
Description: Changes in endometrial thickness between the 3 groups.
Time Frame: Baseline, and Visit 4 (end of study, up to 40 days)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | EGCG Daily Alone. | EGCG With Clomiphene Citrate | EGCG With Letrozole
Number analyzed (Participants) | 13 | 11 | 11
mm | -1.9 (4.3) | 1.4 (2.0) | 0.6 (2.7)
Statistical Analysis 1: Comparison: EGCG Daily Alone. vs EGCG With Clomiphene Citrate vs EGCG With Letrozole; Test type: Superiority; p = 0.146, Kruskal-Wallis

9. Secondary Outcome: Change in Serum Folate Level Between MTHFR677-Wild Type (WT) Group and MTHFR677-Hetero Group
Description: Change in serum folate levels between MTHFR677-Wild Type (WT) group and MTHFR677-Hetero group
Time Frame: Baseline, and Visit 4 (end of study, up to 40 days)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- MTHFR677-Wild Type (WT) Group: MTHFR677-Wild Type (WT) group
- MTHFR677-Hetero Group: MTHFR677-Hetero group
Arm/Group | MTHFR677-Wild Type (WT) Group | MTHFR677-Hetero Group
Number analyzed (Participants) | 13 | 17
ng/mL | -3.2 (4.1) | -2.0 (3.0)
Statistical Analysis 1: Comparison: MTHFR677-Wild Type (WT) Group vs MTHFR677-Hetero Group; Test type: Superiority; p = 0.372, t-test, 2 sided

10. Secondary Outcome: Change in Serum Folate Level Between MTHFR1298-Wild Type (WT) Group and MTHFR1298-Hetero Group
Description: Change in serum folate levels between MTHFR1298-Wild Type (WT) group and MTHFR1298-Hetero group
Time Frame: Baseline, and Visit 4 (end of study, up to 40 days)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- MTHFR1298-Wild Type (WT) Group: MTHFR1298-Wild Type (WT) group
- MTHFR1298-Hetero Group: MTHFR1298-Hetero group
Arm/Group | MTHFR1298-Wild Type (WT) Group | MTHFR1298-Hetero Group
Number analyzed (Participants) | 16 | 14
ng/mL | -1.5 (3.0) | -3.8 (3.7)
Statistical Analysis 1: Comparison: MTHFR1298-Wild Type (WT) Group vs MTHFR1298-Hetero Group; Test type: Superiority; p = 0.07, t-test, 2 sided

11. Secondary Outcome: Change in Serum Folate Level Between DHFR-Wild Type (WT) Group and DHFR-Hetero or Homo Group.
Description: Change in serum folate levels between DHFR-Wild Type (WT) group and DHFR-Hetero or homo group.
Time Frame: Baseline, and Visit 4 (end of study, up to 40 days)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- DHFR-Wild Type (WT) Group: DHFR-Wild Type (WT) group
- DHFR-Hetero or Homo Group.: DHFR-Hetero or homo group.
Arm/Group | DHFR-Wild Type (WT) Group | DHFR-Hetero or Homo Group.
Number analyzed (Participants) | 7 | 23
ng/mL | -3.9 (4.3) | -2.1 (3.2)
Statistical Analysis 1: Comparison: DHFR-Wild Type (WT) Group vs DHFR-Hetero or Homo Group; Test type: Superiority; p = 0.24, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 60 days
Arm/Group | EGCG Daily Alone. | EGCG With Clomiphene Citrate | EGCG With Letrozole
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 2/16 | 4/11 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EGCG Daily Alone. (N=16) | EGCG With Clomiphene Citrate (N=11) | EGCG With Letrozole (N=12)
Abdominal discomfort and loose stool (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Dizziness (General disorders) | 0 | 1 | 0
Facial flushing, muscle ache, and diarrhea after letrozole (General disorders) | 0 | 0 | 1
Greenish discharge (Gastrointestinal disorders) | 0 | 1 | 0
Headaches (General disorders) | 1 | 0 | 0
Insomnia (General disorders) | 0 | 1 | 1
Kidney pain (Renal and urinary disorders) | 0 | 0 | 1
Loose stool (Gastrointestinal disorders) | 0 | 0 | 1
Low mood (General disorders) | 0 | 1 | 0
Migraine after vaccine (Immune system disorders) | 1 | 0 | 0
Nausea with EGCG (Gastrointestinal disorders) | 0 | 1 | 1
Pelvic cramps, dull and intermittent aching after letrozole (General disorders) | 0 | 0 | 1
Vomiting and diarrhea after clomid (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT04177693/Prot_SAP_000.pdf